CLINICAL TRIAL: NCT00072488
Title: Whole-Body MRI in the Evaluation of Pediatric Malignancies
Brief Title: Whole-Body MRI and Conventional Imaging in Detecting Distant Metastases in Young Patients With Solid Tumors or Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000339811; ACRIN-6660; NCT00228761 (obsolete NCT alias)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2007-10

CONDITIONS: Lymphoma; Neuroblastoma; Sarcoma
Keywords: disseminated neuroblastoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma; previously untreated childhood rhabdomyosarcoma; stage I childhood Hodgkin lymphoma; stage I childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood Hodgkin lymphoma; stage II childhood large cell lymphoma; stage II childhood lymphoblastic lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood Hodgkin lymphoma; stage III childhood large cell lymphoma; stage III childhood lymphoblastic lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood Hodgkin lymphoma; stage IV childhood large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; previously treated childhood rhabdomyosarcoma
MeSH Terms: conditions — Lymphoma; Neuroblastoma; Sarcoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: computed tomography
Procedure: magnetic resonance imaging
Procedure: positron emission tomography

SUMMARY:
RATIONALE: New imaging procedures, such as whole-body MRI, may improve the ability to detect metastatic cancer and determine the extent of disease.

PURPOSE: This clinical trial is studying whole-body MRI to see how well it works compared to standard imaging procedures in detecting distant metastases in patients with solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare non-inferior diagnostic performance of whole-body MRI (i.e., combination of turbo short-tau inversion-recovery (STIR) and out-of-phase imaging) vs conventional imaging (i.e., the combination of chest CT scan, scintigraphy [bone, gallium, meta-iodobenzylguanidine (MIBG), or optional fludeoxyglucose F 18 positron emission tomography (FDG-PET)] and abdominal/pelvic CT scan/MRI as indicated) for detecting distant metastases for use in staging common tumors in pediatric patients.

Secondary

* Determine the incremental benefit of adding out-of-phase T1-weighted gradient-recalled echo imaging to turbo STIR for detecting distant disease in these patients.
* Determine, preliminarily, the relative accuracies of FDG-PET, whole-body MRI, and a combination of FDG-PET and whole-body MRI in detecting stage IV disease in these patients.
* Determine the effects of multiple factors, including cancer type, site of primary tumor, and patient age, on diagnostic accuracy of whole-body MRI in these patients.
* Determine the interobserver variability associated with interpreting whole-body MRI exams for detecting distant metastases in these patients.

OUTLINE: This is a multicenter study.

Patients undergo conventional MRI, CT scan, and/or scintigraphy (e.g., bone, meta-iodobenzylguanidine [MIBG], or gallium) and experimental whole-body MRI sequences. Patients may optionally undergo fludeoxyglucose F18 positron emission tomography (FDG-PET).

Patients with a lesion (or lesions) detected on whole-body MRI or FDG-PET at initial staging that are not confirmed by biopsy or other conventional imaging studies at staging repeat standard imaging at 3- to 6-month follow-up.

Patients with an abnormality that is considered highly suspicious for a metastasis or when biopsy proof of that metastasis is obtained receive treatment at the discretion of the treating physician.

Patients are followed annually for 3 years.

PROJECTED ACCRUAL: A total of 226 patients (45 with neuroblastoma, 54 with rhabdomyosarcoma, 27 with other sarcoma, and 100 with lymphoma) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis OR newly diagnosed mass strongly suspected to represent 1 of the following:

  * Rhabdomyosarcoma
  * Ewing's sarcoma family of tumors
  * Neuroblastoma
  * Hodgkin's lymphoma
  * Non-Hodgkin's lymphoma
* All imaging examinations (e.g., CT scan, MRI, or scintigraphy) must be performed within 14 days of each other and within 2 months of any diagnostic or operative procedure

  * Whole body MRI and positron emission tomography (PET) scanning (if PET scan is being done) must be done before treatment
  * Prior CT scan, conventional MRI, bone scintigraphy, gallium scintigraphy, or meta-iodobenzylguanidine (MIBG) scintigraphy performed at outside institutions allowed provided the same technical standards specified in this study were practiced
  * Bone scintigraphy required for patients with neuroblastoma, rhabdomyosarcoma, or other sarcomas
  * Gallium scintigraphy not required in lymphoma patients if PET scan is performed
* No CNS primary tumor

PATIENT CHARACTERISTICS:

Age

* 21 and under

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No active cardiac pacemakers

Other

* Not pregnant or nursing
* No prior malignancy
* No uncontrolled diabetes mellitus (for patients undergoing optional PET)

  * Patients with controlled diabetes mellitus must have a fasting blood glucose no greater than 200 mg/dL
* No contraindications to MRI or CT scan (e.g., intracranial vascular clips)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Prior biopsy or surgery allowed provided no more than 2 months has passed since the procedure

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 226 (Estimated)
Dates: Start 2004-10; Primary Completion 2005-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn J. Siegel, MD, Principal Investigator — Mallinckrodt Institute of Radiology at Washington University Medical Center
Locations (21):
- United States (17):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Riley's Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mallinckrodt Institute of Radiology at Washington University Medical Center, St Louis, Missouri
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- Canada (4):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario